CLINICAL TRIAL: NCT03191019
Title: Design and Evaluation of a Mobile-phone Based Intervention to Support Smoking Cessation Among Chilean Women Aged 18 to 44 Years in the Metropolitan Region
Brief Title: A Mobile-phone Based Intervention to Support Smoking Cessation Among Chilean Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15-349; FONIS SA15I20120 (Other: National Commission for Scientific & Technological Research)
Record Dates: First submitted 2017-06-14; First posted 2017-06-19 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Smoking Cessation
Keywords: Cell phones; Women
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Intervention Model Description: Two-arm, randomized clinical trial of a smoking cessation intervention based on a mobile-phone app. Participants will be randomly assigned to the intervention group or control group, in parallel for the duration of the study (6 months follow-up).
Who Masked: Investigator, Outcomes Assessor
Masking Description: Eligible participants will be randomized to the intervention group or control group using a computerized and automated process. An email will be automatically sent to the participants with the link to download the corresponding version of the mobile-phone app (intervention app or control app). Researchers who will gather data and those who will measure carbon monoxide in exhaled air will be masked to treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile-phone app for smoking cessation (Experimental): The intervention arm will receive a smoking cessation program based on a mobile-phone app. The program contains strategies to support smoking cessation, including motivational messages, tips on stress management, on how to ask support from friends and family, how to use distraction techniques and how to deal with cravings, lapses and early relapse. It also includes a saving calculator, a "help button" which provides extra messages in case of cravings and a "lapse button", which provides advice about what to do if the participant presents lapses or relapse after being abstinent at least 24 hours.
  Interventions: Behavioral: Mobile-phone app for smoking cessation
- Control mobile-phone app (Placebo Comparator): The control arm will receive a mobile-phone app which will send 1 message every two weeks thanking participants for taking part in the study, and encouraging them to stay in the study for the 6 month follow-up period.
  Interventions: Behavioral: Mobile-phone app for smoking cessation

INTERVENTIONS:
Behavioral: Mobile-phone app for smoking cessation — Android App for smoking cessation

SUMMARY:
The purpose of this study is to determine whether a mobile-phone based intervention is effective in supporting smoking cessation among Chilean women

DETAILED DESCRIPTION:
This protocol corresponds to a single-blind, two-arm, randomized clinical trial of a smoking cessation intervention based on a mobile-phone app. Eligible participants are Chilean women from the Metropolitan Region, who smoke daily (at least one cigarette per day) or weekly (at least 7 cigarettes per week), and who are willing to make a quit attempt within one month of enrollment. Study will be advertised on the local radio, primary care centers, smoking cessation services and through social media campaigns. Study information will be available online. Potential participants will be asked to register their interest by sending an email to the study. Research assistants then will contact respondents by phone in order to complete a baseline questionnaire about sociodemographic variables, characteristics of tobacco consumption, and to assess eligibility for the study. Eligible participants will be then randomized to the intervention group or control group using a computerized and automated process, in blocks of 6. A minimization algorithm balancing for Fagerstrom score for nicotine addiction (≤5, >5) will be used. Researchers who will gather data and those who will measure carbon monoxide in exhaled air will be masked to treatment allocation.

Each participant will be emailed the link with either the intervention or the control version of the mobile-phone app. Once participants download the app, they will be asked to provide informed consent by clicking the "accept" or "reject" button in the app.

Participants randomized to the intervention app will be sent motivational and preparatory content for the first two weeks, and they will be asked to set a quit date within 4 weeks from enrollment. The mobile app will send an average of 4 messages per day during the first month after quit date, followed by three messages per week up to the end of the study at month 6.

The intervention program was designed based on current best evidence on strategies to support smoking cessation, and included work of Chilean experts in smoking cessation. The design of the intervention app also included the opinion and preferences of potential participants who participated in focus groups during intervention design. The intervention app includes motivational messages, tips on stress management, on how to ask support from friends and family, how to use distraction techniques and how to deal with cravings, lapses and early relapse.

The intervention app also includes a "help button" which provides extra messages in case of cravings and a "lapse/relapse button", which provides advice about what to do if the participant returned to smoke. The control group will receive a control app which will send 1 message every two weeks thanking participants for taking part in the study, and encouraging them to stay in the study for the 6 month follow-up period. After completing the 6-month follow-up evaluation, the control group will be offered access to the intervention app.

Women will not receive financial compensation for their participation in the study. In order to increase retention, participants in both arms will be told that they would be entered into a lottery for different prizes after answering the 6-month follow-up questionnaire.

For the 4-week, 3-month and 6-month follow-up, a link to an electronic follow-up questionnaire will be emailed to all participants. Reminders will be sent to non responders and if they still do not respond, additional email reminders will be sent. If participants still do not respond, research assistants will call them by phone in order to capture the primary outcome of the study. At 6-month follow-up, participants who reported having quit smoking will be asked to attend to the local primary care center in order to measure carbon monoxide in exhaled air. All measurements will be performed by research assistants who are masked to treatment allocation.

Sample size was calculated based on previous studies. Twenty-eight percent quitting in the intervention group and 13% in the control group was expected. To achieve 90% power with a significance level of P ≤ .05 (2-sided), and including a 20% attrition for the 6 month follow-up evaluation, a sample size of 400 was estimated. In order to take into account that the size effect associated to the intervention could be lesser in Chile than the reported for other countries, investigators defined a 90% power for the sample size calculation.

Investigators plan to conduct analyses for the whole sample and also for subgroups of age (<35 years, ≥35 years), nicotine addiction (Fagerstrom score ≤5, >5), educational level (<8 years, 8-12 years, ≥12 years), and use of other smoking cessation treatments or services during the trial (yes, no).

All statistical analyses for clinical effectiveness will be undertaken on an intention-to-treat basis. For missing observations in the primary outcome, two methods will be used: last value carried forward method and multiple imputation method, as attempts to correct for potential bias caused by missing data.

Analyses for adverse effects outcomes will be performed on a per-protocol basis.

ELIGIBILITY:
Inclusion Criteria:

* Smoker of at least 1 cigarette per day or at least 7 cigarettes per week in the last 6 months
* Willing to make a quit attempt in the next month
* Owns and uses an Android cell phone
* Lives in the Metropolitan Region and has no plans to move in the next year

Exclusion Criteria:

* Severe mental disability or inability to read or answer a telephone survey
* Screening positive for hazardous drinking behavior or active alcohol use disorder

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 309 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2018-07-22 (Actual); Study Completion 2018-11-04 (Actual)

PRIMARY OUTCOMES:
Point prevalence of smoking abstinence at 4 weeks | 4 weeks
  Self-reported no smoking in past 7 days at 4 weeks from quit date

SECONDARY OUTCOMES:
Continuous smoking abstinence at 4 weeks | 4 weeks
  Self-report of continuous abstinence (< 5 cigarettes) at 4 weeks
Point prevalence of smoking abstinence at 3 months | 3 months
  Self-reported no smoking in past 7 days at 3 months from quit date
Continuous smoking abstinence at 3 months | 3 months
  Self-report of continuous abstinence (< 5 cigarettes) at 3 months
Point prevalence of smoking abstinence at 6 months | 6 months
  Self-reported no smoking in past 7 days at 6 months from quit date
Biochemically verified continuous smoking abstinence at 6 months | 6 months
  Self-report of continuous abstinence (< 5 cigarettes) and passed carbon monoxide validation at 6 months
Quit attempts | 6 months
  Mean number of quit attempts since taking part in the study
Use of other smoking cessation services | 6 months
  Number of uses of other smoking cessation services since taking part in the study
Number of cigarettes smoked per day or weekly at 6 months | 6 months
  Mean number of cigarettes smoked per day or weekly among participants still smoking at 6 months
Adverse events vehicle crashes | 6 months
  Involvement in any vehicle crashes since taking part in the study
Adverse events hand injury | 6 months
  Repetitive strain injury of the hand related to use of mobile-phone since taking part in the study

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Bambs, Study Director — Pontificia Universidad Catolica de Chile
Locations (1):
- Centro de Salud Familiar Madre Teresa de Calcuta, Santiago, Other (Non U.s.), Chile

IPD SHARING:
Plan to Share IPD: No